CLINICAL TRIAL: NCT02359890
Title: Prospective Safety Assessment of the THERMOCOOL® SMARTTOUCH® SF Family of Contact Force Sensing Catheters for the Radiofrequency Ablation Treatment of Drug Refractory Symptomatic Paroxysmal Atrial Fibrillation
Brief Title: SMART-SF Radiofrequency Ablation Safety Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMART-SF; STSF-162 (Other: BiosenseWebster)
Record Dates: First submitted 2015-02-03; First posted 2015-02-10 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: Interventional; Radiofrequency ablation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Group (Experimental): Pulmonary vein isolation by RF ablation treatment with the THERMOCOOL® SMARTTOUCH® SF family of contact force sensing catheters (study device)
  Interventions: Device: THERMOCOOL® SMARTTOUCH® (RF ablation treatment)

INTERVENTIONS:
Device: THERMOCOOL® SMARTTOUCH® (RF ablation treatment) — Radiofrequency Ablation Treatment
  Other Names: Pulmonary vein isolation

SUMMARY:
This is a prospective safety assessment of the study device during radiofrequency (RF) ablation treatment of patients with drug refractory symptomatic atrial fibrillation (SMART-SF).

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the safety of the study device in the treatment of drug refractory symptomatic paroxysmal atrial fibrillation (PAF) during standard electrophysiology mapping and RF ablation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal atrial fibrillation (AF) who have had at least one AF episode electrocardiographically documented within one (1) year prior to enrollment and a physician's note indicating recurrent, self-terminating AF. Electrocardiographic documentation may include, but is not limited to, electrocardiogram (ECG), transtelephonic monitor (TTM), Holter monitor (HM), or telemetry strip
* Failed at least one antiarrhythmic drug (AAD) (class I or III, or atrioventricular (AV) nodal blocking agents such as beta blockers and calcium channel blockers) as evidenced by recurrent symptomatic AF, or intolerable to the AAD
* Age 18 years or older

Exclusion Criteria:

* Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* Previous surgical or catheter ablation for atrial fibrillation
* Amiodarone at any time during the past 3 months
* Any percutaneous coronary intervention (PCI), cardiac surgery, or valvular cardiac surgical or percutaneous procedure (e.g., ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve) within the past 2 months
* Any carotid stenting or endarterectomy
* Coronary artery bypass graft (CABG) surgery within the past 6 months
* AF episodes lasting >7 days
* Documented left atrial (LA) thrombus on imaging
* LA size >50 mm
* Left ventricular ejection fraction (LVEF) < 40%
* Contraindication to anticoagulation (heparin or warfarin)
* History of blood clotting or bleeding abnormalities
* MI within the past 2 months
* Documented thromboembolic event (including transient ischemic attack (TIA)) within the past 12 months
* Rheumatic Heart Disease
* Uncontrolled heart failure or New York Heart Association (NYHA) function class III or IV
* Awaiting cardiac transplantation or other cardiac surgery within the next 12 months
* Unstable angina
* Acute illness or active systemic infection or sepsis
* Diagnosed atrial myxoma
* Presence of implanted implantable cardioverter defibrillator (ICD)
* Significant pulmonary disease, (eg, restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
* Women who are pregnant (as evidenced by pregnancy test if pre-menopausal)
* Enrollment in an investigational study evaluating another device, biologic, or drug
* Presence of intramural thrombus, tumor or other abnormality that precludes vascular access, or manipulation of the catheter
* Presence of a condition that precludes vascular access
* Life expectancy or other disease processes likely to limit survival to less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2016-11-08 (Actual)

REFERENCES:
- [Background] Natale A, Reddy VY, Monir G, Wilber DJ, Lindsay BD, McElderry HT, Kantipudi C, Mansour MC, Melby DP, Packer DL, Nakagawa H, Zhang B, Stagg RB, Boo LM, Marchlinski FE. Paroxysmal AF catheter ablation with a contact force sensing catheter: results of the prospective, multicenter SMART-AF trial. J Am Coll Cardiol. 2014 Aug 19;64(7):647-56. doi: 10.1016/j.jacc.2014.04.072. PMID 25125294
- [Background] Oza SR, Hunter TD, Biviano AB, Dandamudi G, Herweg B, Patel AM, Pollak SJ, Wang H, Fishel RS. Acute safety of an open-irrigated ablation catheter with 56-hole porous tip for radiofrequency ablation of paroxysmal atrial fibrillation: analysis from 2 observational registry studies. J Cardiovasc Electrophysiol. 2014 Aug;25(8):852-858. doi: 10.1111/jce.12403. Epub 2014 Apr 9. PMID 24602038
- See also: Sponsor website — http://BiosenseWebster.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 165 subjects at 17 clinical sites in the U.S. over approximately 5 months. The first subject was enrolled on March 30, 2015 and the last subject was enrolled on September 9, 2015. The last ablation procedure was on September 17, 2015. The last 1-month follow-up visit occurred on November 3, 2015.
Groups:
- THERMOCOOL SMARTTOUCH® SF Family of Catheters: Pulmonary vein isolation by radiofrequency (RF) ablation treatment with the THERMOCOOL® SMARTTOUCH® SF family of contact force sensing catheters (study device)
Period: Overall Study
Arm/Group | THERMOCOOL SMARTTOUCH® SF Family of Catheters
Started | 165 (Patients who enrolled in the study are those who signed informed consent forms.)
Safety Population | 159 (Enrolled subjects who had the study catheter inserted)
mITT Population | 155 (Enrolled subjects who met the inclusion/exclusion criteria and had the study catheter inserted)
Per-Protocol (PP) Population | 155 (Subjects part of mITT population who had undergone RF ablation.)
Completed | 155
Not Completed | 10
Not completed — Not meeting eligibility | 4
Not completed — Never treated with study catheter | 6

BASELINE CHARACTERISTICS:
Population: Enrolled patients who had baseline data available
Arm/Group | THERMOCOOL SMARTTOUCH® SF Family of Catheters
Number analyzed (Participants) | 164
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age (Years) | 62.7 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 155
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 159
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Early Onset Primary Adverse Events
Description: Early onset is defined as within 7 days of the atrial fibrillation (AF) ablation procedure. Primary adverse events (AE) include Death, Myocardial infarction (MI), Pulmonary vein (PV) stenosis, Diaphragmatic paralysis, Atrio-esophageal fistula, Transient Ischemic Attack (TIA), Stroke / Cerebrovascular accident (CVA), Thromboembolism, Pericarditis, Cardiac Tamponade / Perforation, Pneumothorax, Major Vascular Access Complications / Bleeding, Pulmonary edema (Respiratory Insufficiency), and Heart block.
Time Frame: Seven days post ablation procedure
Population: The modified intent-to-treat (mITT) population was used, which consisted of enrolled subjects who met the eligibility criteria and had the study catheter inserted.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- THERMOCOOL SMARTTOUCH® SF Catheters: Pulmonary vein isolation by radiofrequency (RF) ablation treatment with the THERMOCOOL® SMARTTOUCH® SF family of contact force sensing catheters (study device)
Arm/Group | THERMOCOOL SMARTTOUCH® SF Catheters
Number analyzed (Participants) | 155
Percentage of participants | 2.6 [0.7 to 6.5]
Statistical Analysis 1: Comparison: THERMOCOOL SMARTTOUCH® SF Catheters; Test type: Superiority or Other; Percentage of participants with events = 2.6, 95% CI 2-sided [0.7 to 6.5] — The 2-sided 95% confidence interval is derived using the exact Clopper-Pearson interval

2. Secondary Outcome: Percentage of Participants With Non-Primary Serious Adverse Events (SAEs)
Description: This secondary safety endpoint includes non-primary serious adverse events (SAEs) within 7 days post-procedure and serious adverse events from 8 days to 30 days post-procedure
Time Frame: Up to 30 days post Procedure
Population: Safety Population (SP), which is defined as the enrolled subjects who had the study catheter inserted.
Measure: Number; unit: Percentage of Participants
Arm/Group | THERMOCOOL SMARTTOUCH® SF Catheters
Number analyzed (Participants) | 159
Percentage of Participants
  Patients with SAE within 7 days post procedure | 3.1
  Patients with SAE during 8-30 days post-procedure | 0.6

3. Secondary Outcome: Percentage of Participants With Acute Success
Description: Acute success is defined as confirmation of entrance block in all Pulmonary veins (PV).
Time Frame: End of procedure
Population: Safety Population (SP), which is defined as the enrolled subjects who had the study catheter inserted.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | THERMOCOOL SMARTTOUCH® SF Catheters
Number analyzed (Participants) | 159
Percentage of participants | 96.2 [92.0 to 98.6]
Statistical Analysis 1: Comparison: THERMOCOOL SMARTTOUCH® SF Catheters; Test type: Superiority or Other; Percentage of patient with acute success = 96.2, 95% CI 2-sided [92.0 to 98.6] — The 2-sided 95% confidence interval is derived using the exact Clopper-Pearson interval

4. Secondary Outcome: Effectiveness Endpoint: Freedom From Documented Atrial Fibrillation (AF)/Atrial Tachycardia (AT)/Atrial Flutter (AFL)
Description: The freedom from documented AF/AT/AFL based on electrocardiographic data
Time Frame: 12 months
Population: Effectiveness per Protocol Population, which is defined as enrolled subjects who underwent RF ablation procedure with study catheter and completed the 12 month visit.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | THERMOCOOL SMARTTOUCH® SF Catheters
Number analyzed (Participants) | 76
Percentage of Participants | 75 [65.5 to 83.0]

ADVERSE EVENTS:
Time Frame: 30 days post procedure
Arm/Group | THERMOCOOL SMARTTOUCH® SF Family of Catheters
Serious Adverse Events (participants affected / at risk) | 9/159
Other Adverse Events (participants affected / at risk) | 31/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL SMARTTOUCH® SF Family of Catheters (N=159)
Sepsis due to urinary tract and upper respiratory infection (Infections and infestations) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization due to transient neurological symptoms (Eye disorders) | 1 (1)
Abdominal pain/nausea/constipation (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 1 (1)
Septic shock due to pneumonia with abscess (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 2 (2)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Thromboembolism (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL SMARTTOUCH® SF Family of Catheters (N=159)
Groin hematoma (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
UTI (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Globus feeling in pharynx (General disorders) | 1 (1)
Chest pressure (General disorders) | 1 (1)
Catheter site edema (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Radiating chest pain (General disorders) | 2 (2)
Chest pain/discomfort (General disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 4 (4)
Atrial Tachycardia (Cardiac disorders) | 1 (1)
Paroxysmal SVT (Cardiac disorders) | 1 (1)
Atypical left atrial flutter (Cardiac disorders) | 1 (1)
Shock (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Numbness in feet (Nervous system disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Injury, poisoning and procedural complications) | 1 (1)
Poison ivy exposure (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Additional data pertaining to this study expected to be submitted in August 2018. Re-monitoring of safety event data is in progress.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.